CLINICAL TRIAL: NCT06271837
Title: A Phase II, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Trastuzumab Deruxtecan (T-DXd, DS-8201a) as Monotherapy or in Combination With Anti-cancer Agents for the Treatment of Patients With Selected HER2-expressing Tumors (DESTINY PanTumor03)
Brief Title: A Study of T-DXd as Monotherapy or in Combination With Anti-cancer Agents in Patients With Selected HER2-expressing Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D781AC00001
Record Dates: First submitted 2024-01-19; First posted 2024-02-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors (Excluding Gastric Cancer and Breast Cancer)
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Bevacizumab

STUDY DESIGN:
Masking Description: This study is Open-Label Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): HER2 IHC 3+ solid tumors (excluding breast and gastric cancer)
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort A (Experimental): HER2 IHC 2+ solid tumors (excluding breast and gastric cancer)
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort B (Experimental): HER2 IHC 1+ gynecologic cancers
  Interventions: Drug: Trastuzumab deruxtecan
- Part 3 (Experimental): HER2 IHC 3+ or 2+ cervical cancer
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan by intravenous infusion
  Other Names: DS-8201a; T-DXd
Drug: Bevacizumab — Bevacizumab by intravenous infusion
  Arms: Part 3

SUMMARY:
This is an open-label, multicenter, Phase II study to evaluate the efficacy and safety of trastuzumab deruxtecan as monotherapy or in combination with anti-cancer agents for the treatment in locally advanced, unresectable, or metastatic patients with selected HER2-expressing solid tumors which are not eligible for curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Locally advanced, unresectable, or metastatic solid tumors based on most recent imaging.
* HER2 expression.
* ECOG performance status of 0-1.
* Must provide an adequate FFPE tumor sample to centrally determine HER2 status and other correlatives.
* Has measurable target disease assessed by the investigator based on RECIST 1.1.
* Adequate organ function and bone marrow within 14 days before enrollment.
* Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.
* Provision of signed and dated written ICF prior to mandatory study-specific procedures, sampling, or analyses.
* Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner.

Exclusion Criteria:

* Primary diagnosis of adenocarcinoma of the breast, adenocarcinoma of the gastric body or gastroesophageal junction.
* Has substance abuse or any other medical conditions that may interfere with the patient's participation in the clinical study or evaluation of the clinical study results.
* A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and concentrated ascites reinfusion therapy.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated.
* Has unresolved toxicities from previous anti cancer therapy.
* Has any spinal cord compression, leptomeningeal disease, or clinically active CNS metastases.
* Uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals, or active infection including tuberculosis.
* Active primary immunodeficiency, known uncontrolled active HIV infection, or active Hepatitis B or C infection.
* Protocol-defined inadequate cardiac function.
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has a concomitant medical condition that would increase the risk of toxicity in the opinion of the investigator.
* Anti cancer chemotherapy without an adequate treatment washout period prior to enrollment.
* Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
* Known allergy or hypersensitivity to study treatment or any excipients of the product or other mAbs.
* Involvement in the planning and/or conduct of the study.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Previous enrollment in the present study. Concurrent enrollment in another therapeutic clinical study (excluding observational studies).
* For females only: Currently pregnant or breast feeding, or who are planning to become pregnant.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | An average of approximately 12 months
  Confirmed ORR is the proportion of patients who have a confirmed complete response or confirmed partial response per RECIST 1.1.

SECONDARY OUTCOMES:
Duration of Response (DoR) | An average of approximately 12 months
  DoR is defined as the time from the date of first documented response until the date of documented progression (per RECIST 1.1) or death in the absence of disease progression.
Disease control rate (DCR) | An average of approximately 12 months
  The DCR is defined as the percentage of patients who have a confirmed complete response (CR) or partial response (PR) or stable disease (SD) per RECIST 1.1.
Confirmed best objective response (BOR) | An average of approximately 12 months
  BOR is a patient's best response during their participation in the study up until RECIST 1.1-defined progression or the last evaluable assessment in the absence of RECIST 1.1-defined progression.
Progression-free survival (PFS) | An average of approximately 12 months
  PFS is defined as the time from the date of enrollment until the date of objective progressive disease (PD) per RECIST 1.1 or death.
Overall survival (OS) | An average of approximately 12 months
  OS is defined as the time from the date of enrollment until death due to any cause.
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | An average of approximately 12 months
  The grading scales found in the revised NCI CTCAE v5.0 will be utilized for all events.
Pharmacokinetics (PK) of T-DXd | An average of approximately 12 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for T-DXd, total anti-HER2 antibody and MAAA-1181a.
Immunogenicity of T-DXd | An average of approximately 12 months
  Incidence of anti-drug antibodies against T-DXd in serum at each time point.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongyang
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Lishui
  - Research Site, Nanchang
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home